CLINICAL TRIAL: NCT04209023
Title: The Use of Navigated Transcranial Magnetic Stimulation (nTMS) in the Inhibition of Neurofunctional Regions of Interest
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending end of COVID-19 pandemic
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 20193155
Record Dates: First submitted 2019-12-19; First posted 2019-12-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Brain Tumor; Surgery
Keywords: glioma; transcranial magnetic stimulation; neurofunctional inhibition; fMRI verification
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Selected patients will undergo 1 session of TMS treatment to include a non-TMS baseline task and a TMS testing task. The baseline and the testing task are the self-same task. The baseline test demonstrates patient comprehension of instructions, as well as a baseline of task performance for comparison analysis. The TMS test will include the self-same task that may be randomized in terms of order of stimulus presentation. Each component--the baseline and the TMS task--will have a duration of 10 minutes, for a total intervention time of 20 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- navigated TMS (Experimental): All patients are required to have an advanced MRI of the brain including a structural T1, volume measurements of various brain regions, ASL, and BOLD sequences. Patients will also undergo an in-scanner task designed to activate key neurofunctional regions of interest; these areas will provide the cerebral coordinates to be validated by TMS.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Individual pulses (100% motor threshold intensity, continuous temperature of 24 degrees C) will be delivered upon the presentation of the stimulus or the verbal command for the language tasks. Two research coordinators will perform the intervention, with one coordinator presenting the stimulus/giving commands, and the other positioning the TMS coil and delivering the individual pulse or pulse trains. The stimulus presentation will last for a duration of 1 second, in conjunction with the time-course of the pulse's disruption. One or both research coordinators must track the successful or unsuccessful inhibition of task completion for each trial. The number of trials may vary depending on task and region-of-interest; however the intervention is not to exceed a total of 20 minutes.

SUMMARY:
The purpose of this study is to investigate the efficacy of task inhibition during TMS to confirm brain region localization. This study could provide an effective pathway for neurofunctional landmark confirmation that may be useful in a number of treatment modalities and medical considerations.

DETAILED DESCRIPTION:
Selected patients will undergo 1 session of TMS treatment to include a non-TMS baseline task and a TMS testing task. The baseline and the testing task are the self-same task. The baseline test demonstrates patient comprehension of instructions, as well as a baseline of task performance for comparison analysis. The TMS test will include the self-same task that may be randomized in terms of order of stimulus presentation. Each component--the baseline and the TMS task--will have a duration of 10 minutes, for a total intervention time of 20 minutes.

Individual pulses (100% motor threshold intensity, continuous temperature of 24-C) will be delivered upon the presentation of the stimulus or the verbal command for the language tasks. For the motor area, intermittent pulses will be delivered during random finger-tapping. Two research coordinators will perform the intervention, with one coordinator presenting the stimulus/giving commands, and the other positioning the TMS coil and delivering the individual pulse or pulse trains. For the language tasks, both research coordinators need to be well-harmonized: as one coordinator presents the stimulus, the other must simultaneously administer the pulse. The stimulus presentation will last for a duration of 1 second, in conjunction with the time-course of the pulse's disruption. One or both research coordinators must track the successful or unsuccessful inhibition of task completion for each trial. For example, if the patient was able to correctly name all but one picture during TMS, then task inhibition occurred in 1 out of 20 trials, suggesting a failure in the neuronavigation of Broca's area. The number of trials may vary depending on task and region-of-interest; however the intervention is not to exceed a total of 20 minutes. Upon conclusion of the TMS session, the patient will discuss the outcome with the treating physician and follow-on procedures will be scheduled. Patients will not need to undergo a post-treatment MRI, as the MRI scans are functioning as a technique for neuronavigation for precise targeting.

The safety of this protocol will be closely monitored and data will be used to determine whether any significant safety issues exist when using TMS therapy. Adverse events will be noted whenever they occur but will be recorded at the time of the TMS procedure.

All patients will have a thorough discussion to obtain informed consent. Additional meetings with the physicians will further clarify the nature of the study, reasons for transcranial magnetic stimulation, and the possible risks involved. The nature of this study does not require randomization, but rather attempts to isolate adverse and advantageous events should they occur.

ELIGIBILITY:
Inclusion Criteria:

* Indicated need for neuronavigated TMS (e.g. in the case of surgical resection of tumors affecting functional areas such as Broca's, Wenicke's, or motor cortex) which may be optimized by confirmation of specified brain regions using TMS.
* At least 18 years of age
* Must be willing to comply with the study protocol
* English Proficiency

Exclusion Criteria:

* Not English Proficient
* Advanced stages of any terminal illness or any active cancer that requires chemotherapy
* History of epilepsy or seizure, or history of such in first degree relative
* An increased risk of seizure for any reason
* Stents in the neck or brain
* Aneurysm clips or coils
* Metal devices/objects in or near the head
* Metallic implants near the ears and eyes
* Facial tattoos with metallic or magnetic-sensitive ink
* Hepatic impairment
* Significant cytopenia
* Cardiovascular, cerebrovascular, and peripheral vascular arterial thrombosis
* Neurodegenerative diseases
* Myeloproliferative disorders
* Women who are pregnant, may become pregnant, or are breastfeeding
* Subjects unable to give informed consent or in vulnerable categories, such as prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-12-16 (Estimated); Primary Completion 2024-12-18 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
TEST FOR BROCA'S AREA (ONLY): Confrontation Naming Task | Baseline prior to TMS administration
  A slideshow of common pictures will be presented one by one; this 20 minute task will establish baseline performance and comprehension of instructions.
TEST FOR BROCA'S AREA (ONLY): Confrontation Naming Task | Testing during TMS administration
  A slideshow of common pictures will be presented one by one.
TEST FOR WERNICKE'S AREA (ONLY): Testing Compliance to Verbalized Commands | Baseline prior to TMS administration
  The following verbal instructions will be given to establish baseline performance and comprehension of instructions:
  "When I say "tongue", stick out your tongue. Do you understand the instructions?" (Receive verbal confirmation of comprehension) "Tongue." "When I say hand, raise your hand. Do you understand the instructions?" (Receive verbal confirmation of comprehension) "Hand." "When I say foot, lift your foot. Do you understand the instructions?" (Receive verbal confirmation of comprehension) "Foot.
  *repeat for duration of baseline test*
TEST FOR WERNICKE'S AREA (ONLY): Testing Compliance to Verbalized Commands | Testing during TMS administration
  The following verbal instructions will be given during the test phase
  Upon each command, a pulse will be delivered.
  "Tongue." (pulse delivered) "Hand." (pulse delivered) "Tongue." (pulse delivered) "Tongue." (pulse delivered) "Foot." (pulse delivered) "Hand." (pulse delivered) "Foot." (pulse delivered)
  *repeat for duration of TMS test*
TEST FOR MOTOR AREA (ONLY): Testing for Finger Tapping Inhibition | Testing during TMS administration
  (A brief baseline measure (30 seconds) for patient to randomly tap fingers wherein no pulses are delivered).

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — The Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Data from this study will not be made publicly available due to ethical and privacy concerns. Anonymized data will be available upon reasonable request from any qualified investigator.

REFERENCES:
- [Background] Cordes D, Haughton VM, Arfanakis K, Wendt GJ, Turski PA, Moritz CH, Quigley MA, Meyerand ME. Mapping functionally related regions of brain with functional connectivity MR imaging. AJNR Am J Neuroradiol. 2000 Oct;21(9):1636-44. PMID 11039342
- [Background] Kannurpatti SS, Rypma B, Biswal BB. Prediction of Task-Related BOLD fMRI with Amplitude Signatures of Resting-State fMRI. Front Syst Neurosci. 2012 Mar 6;6:7. doi: 10.3389/fnsys.2012.00007. eCollection 2012. PMID 22408609
- [Background] Kim CH, Kim JH, Chung CK, Kim JS, Lee JM, Lee SK. Localization of Broca's Area Using Functional MR Imaging: Quantitative Evaluation of Paradigms. J Korean Neurosurg Soc. 2009 Apr;45(4):219-23. doi: 10.3340/jkns.2009.45.4.219. Epub 2009 Apr 30. PMID 19444347
- [Background] Miller GA, Crocker LD, Spielberg JM, Infantolino ZP, Heller W. Issues in localization of brain function: The case of lateralized frontal cortex in cognition, emotion, and psychopathology. Front Integr Neurosci. 2013 Jan 30;7:2. doi: 10.3389/fnint.2013.00002. eCollection 2013. PMID 23386814
- [Background] Rossini PM, Barker AT, Berardelli A, Caramia MD, Caruso G, Cracco RQ, Dimitrijevic MR, Hallett M, Katayama Y, Lucking CH, et al. Non-invasive electrical and magnetic stimulation of the brain, spinal cord and roots: basic principles and procedures for routine clinical application. Report of an IFCN committee. Electroencephalogr Clin Neurophysiol. 1994 Aug;91(2):79-92. doi: 10.1016/0013-4694(94)90029-9. No abstract available. PMID 7519144
- [Background] Ugurbil K, Toth L, Kim DS. How accurate is magnetic resonance imaging of brain function? Trends Neurosci. 2003 Feb;26(2):108-14. doi: 10.1016/S0166-2236(02)00039-5. PMID 12536134
- [Background] Walsh V, Cowey A. Transcranial magnetic stimulation and cognitive neuroscience. Nat Rev Neurosci. 2000 Oct;1(1):73-9. doi: 10.1038/35036239. PMID 11252771